CLINICAL TRIAL: NCT05520918
Title: Clinical Demonstration of a Novel Parameter LIT/N That Predicts Survival in COVID-19 ICU Patients
Brief Title: A Novel Parameter LIT/N That Predicts Survival in COVID-19 ICU Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Collaborators: Oxford MediStress (Unknown)
Responsible Party: Principal Investigator, Nazlıhan Boyacı Dündar, principle invastigator, Gazi University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: GaziUtipNBDundar001
Record Dates: First submitted 2022-08-25; First posted 2022-08-30 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: COVID-19 Pneumonia
Keywords: COVID-19 Pneumonia; ROS; cellular dysfunction of neutrophils

STUDY DESIGN:
Intervention Model Description: Two parallel groups enrolled for baseline LIT scores, that are healthy subjects and COVID-19 pneumonia patients.
  The sequential LIT score were recorded for COVID-19 pneumonia patients during ICU length.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COVID-19 pneumonia patients (Other): sequential LIT was performed to this patient group
  Interventions: Diagnostic Test: the LIT test

INTERVENTIONS:
Diagnostic Test: the LIT test — The retained functional capacity of leukocytes (primarily neutrophils) to produce ROS in response to PMA in whole blood samples could provide a rapid 10-minute detection method for objectively determining onset or occurrence of severe COVID-19 and monitoring progression and treatment of COVID-19.

SUMMARY:
A brisk immune response can clear a pathogen but can cause extensive collateral damage to the host. It is known that coronavirus disease 2019 (COVID-19) infection triggers a multi system inflammatory disorder which can lead to a spectrum of clinical symptoms (Dhama et al. 2020). Severely ill patients maintain a sustained profile of high pro-inflammatory cytokines, (Lucas et al. 2020). Approximately 20% of patients display acute multi-system failure, including acute respiratory distress syndrome (ARDS), accompanied by an intense inflammatory process, which is life-threatening (Wang et al. 2020; Wu et al. 2020; Yang et al. 2020). However, in severe COVID-19, the lymphocyte count decreases progressively, while the neutrophil count gradually increases (Li et al. 2020). To date, four meta-analyses have reported that patients with severe COVID-19 infection have a higher Neutrophil/Lymphocyte ratio (NLR) than those with non-severe COVID-19 infection (Zheng et al. 2020, Chan & Rout. 2020; Ghahramani et al. 2020; Lagunas-Rangel et al. 2020). There is no absolute reported objective threshold level for when NLR progresses from near normal through moderate to severe. An objective marker of cellular dysfunction of neutrophils would be a helpful tool for the clinician in monitoring changes to the patient status and to determine if interventions are having positive effect.

DETAILED DESCRIPTION:
Detailed Description:

It is known that COVID-19 infection triggers a multi system inflammatory disorder which can lead to a spectrum of clinical symptoms (Dhama et al. 2020). Approximately 20% of patients display acute multi-system failure, including ARDS, accompanied by an intense inflammatory process, which is life-threatening (Wang et al. 2020; Wu et al. 2020; Yang et al. 2020). However, in severe COVID-19, the lymphocyte count decreases progressively, while the neutrophil count gradually increases (Li et al. 2020). To date, four meta-analyses have reported that patients with severe COVID-19 infection have a higher NLR than those with non-severe COVID-19 infection (Zheng et al. 2020, Chan & Rout. 2020; Ghahramani et al. 2020; Lagunas-Rangel et al. 2020). There is no absolute reported objective threshold level for when NLR progresses from near normal through moderate to severe.

Neutrophils operate using a number of different mechanisms including chemotaxis, phagocytosis, release of reactive oxygen species (ROS), and granular proteins and the production and liberation of cytokines (Selder et al. 2017; Hellebrekers et al. 2018). Neutrophils are subjected to complex environmental regulation and this can result in significant differences in the production of ROS (Panday et al. 2015 and Nguyen et al. 2017). Veenith and et all have previously demonstrated that ROS production in COVID-19 is dysfunctional (Veenith et al 2022, publishing process). Despite the immense number of studies providing evidence of a dysregulated in vivo innate immune response in some COVID-19 patients, it became apparent that measurement of retained functional capacity of leukocytes (primarily neutrophils) to produce ROS in response to phorbol-12-myristate-13-acetate (PMA) in whole blood samples could provide a rapid 10-minute detection method for objectively determining onset or occurrence of severe COVID-19 and monitoring progression and treatment of COVID-19. A predictive mathematical model would aid the early diagnosis and treatment of COVID-19 and allow clinicians to prioritise patients. Therefore the analysis of the ROS production in response to PMA in COVID-19 pneumonia comparison with healthy subjects may reveal this hypothesis.

Method:

The study was conducted with ethical committee approval in the Intensive Care Unit (ICU) Hospital The patient population consisted of patients who were admitted to the ICU due to COVID-19 pneumonia; the healthy volunteer population consisted of healthcare workers from the hospital. Analysis was performed on clinical samples or via finger-prick assay from healthy volunteers. ROS production in response to PMA was analysed within 30 minutes of collection. Diagnosis of COVID status was confirmed using polymerase chain reaction (PCR) test. Together with a range of conventional haematological tests and clinical observations, the LIT test was performed every day or every other day until death or discharge from the ICU.

Data collection:

Patients were followed from their admission to ICU up to the day of exitus or ICU discharge. All data were prospectively collected on standardized study forms. Data variables collected on admission included the demographic characteristics, diagnosis, comorbidities, date of PCR test positivity, symptoms of COVID-19, severity of COVID-19 (according to world health organisation (WHO) classification), type of treatment, use of ventilation and ventilation type, partial arterial oxygen pressure/inspired oxygen fraction (PaO2/FiO2) ratio , use of antibiotics, C reactive protein (CRP), neutrophil count, total leukocyte count. On admission, severity of the patient was evaluated with APACHE II and severity of organ failure assessment (SOFA) score. During ICU stay, patients were assessed for the development of sepsis or septic shock. The vital signs on the day of LIT test was performed were also recorded. The Intensive care unit outcome parameters such as duration of mechanical ventilation, length of ICU stay, length of hospitalization and mortality were also evaluated. The CRP, neutrophil count and total leukocyte count were performed on the day of LIT test was performed of the healthy volunteers.

Measurements of ROS production by luminometer:

ROS production was measured according to the method previously described [25-27]. Briefly, 10μl samples of freshly obtained blood (obtained by finger prick or venepuncture) was added to 100 microlitres phosphate buffered saline (PBS) containing phorbol 12-myristate 13-acetate (PMA; Sigma) and luminol. The solution was incubated for 10 minutes at 37.5 °C. Chemiluminescence was quantified after 10 minutes using 3MTM handheld luminometer (Clean-Trace, NG3) in relative light units (RLU) . LIT scores as a correlate of neutrophil function for each patient (sampled every day or every other day) and each healthy volunteer (sampled only once) were plotted.

Abnormally high (hyperproduction) or low (hypoproduction) ROS generation was associated with adverse clinical outcomes. This raises the possibility of LIT™/neutrophil-count ratio, (LIT/N), being used as a predictive clinical tool.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COVID-19 pneumonia
* Patients admitted to the ICU due to this clinical diagnosis

Exclusion Criteria:

* Patients who died within 24 hours in the ICU
* Patients who admitted to ICU due to any reason of without COVID-19 pneumonia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
The difference of the LIT scores between COVID-19 pneumonia patients and healthy control | LIT scores of COVID-19 pneumonia patients on the day of ICU admission and a single value of one day in healthy controls
  Comparison of ROS production (LIT scores) between COVID-19 pneumonia patients and volunteer cohorts

SECONDARY OUTCOMES:
The mortality of COVID-19 pneumonia patients | the LIT test was performed every day or every other day until the date of death or discharge from the ICU was occured, assesed up to 6 weeks
  Comparison of LIT scores obtained by repeated measurements in patients with COVID-19 pneumonia in dead and surviving patients

CONTACTS AND LOCATIONS:
Overall Officials: Nazlıhan Boyacı Dündar, assoc. prof, Principal Investigator — principle investigator
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arcanjo A, Logullo J, Menezes CCB, de Souza Carvalho Giangiarulo TC, Dos Reis MC, de Castro GMM, da Silva Fontes Y, Todeschini AR, Freire-de-Lima L, Decote-Ricardo D, Ferreira-Pereira A, Freire-de-Lima CG, Barroso SPC, Takiya C, Conceicao-Silva F, Savino W, Morrot A. The emerging role of neutrophil extracellular traps in severe acute respiratory syndrome coronavirus 2 (COVID-19). Sci Rep. 2020 Nov 12;10(1):19630. doi: 10.1038/s41598-020-76781-0. PMID 33184506
- [Background] Cecchini R, Cecchini AL. SARS-CoV-2 infection pathogenesis is related to oxidative stress as a response to aggression. Med Hypotheses. 2020 Oct;143:110102. doi: 10.1016/j.mehy.2020.110102. Epub 2020 Jul 13. PMID 32721799
- [Background] Ghahramani S, Tabrizi R, Lankarani KB, Kashani SMA, Rezaei S, Zeidi N, Akbari M, Heydari ST, Akbari H, Nowrouzi-Sohrabi P, Ahmadizar F. Laboratory features of severe vs. non-severe COVID-19 patients in Asian populations: a systematic review and meta-analysis. Eur J Med Res. 2020 Aug 3;25(1):30. doi: 10.1186/s40001-020-00432-3. PMID 32746929
- [Background] Lagunas-Rangel FA. Neutrophil-to-lymphocyte ratio and lymphocyte-to-C-reactive protein ratio in patients with severe coronavirus disease 2019 (COVID-19): A meta-analysis. J Med Virol. 2020 Oct;92(10):1733-1734. doi: 10.1002/jmv.25819. Epub 2020 Apr 8. No abstract available. PMID 32242950